CLINICAL TRIAL: NCT05297162
Title: Diagnostic Performance and Clinical Impact of PSMA PET/CT vs. mpMRI in Patients With a High Suspicion of Prostate Cancer and Previously Negative Biopsy: a Head to Head, Parallel, Prospective Trial (PROSPET-BX)."
Brief Title: PSMA PET/CT vs. mpMRI in Patients With a High Suspicion of Prostate Cancer: a Head to Head, Parallel, Prospective Trial
Acronym: PROSPET-BX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3131; GR-2018-12366240 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2021-11-23; First posted 2022-03-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
Keywords: PSMA PET/CT; Primary Diagnosis; multiparametric MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA PET/TRUS (trans-rectal or trans-perineal) fusion biopsy (Experimental): Single-arm case-control imaging trial designed to compare in parallel PSMA PET/TRUS (trans-rectal or trans-perineal) fusion biopsy ("experimental test") with mpMRI/TRUS fusion prostate biopsy ("standard test") in men suspected for PCa after at least one negative biopsy.
  Interventions: Diagnostic Test: PSMA PET/TRUS (trans-rectal or trans-perineal) fusion biopsy

INTERVENTIONS:
Diagnostic Test: PSMA PET/TRUS (trans-rectal or trans-perineal) fusion biopsy — The prostate profile and ROIs will be drawn on PSMA PET and mpMRI and fused in real time with the TRUS image stack during biopsy. Biopsies, transrectal or transperineal according to lesion site, will be performed with patients in the dorsal lithotomy position, under antibiotic prophylaxis and local anesthesia, using 3D triplane transrectal ultrasound system (BK Medical, Analogic Ultrasound Group, Pro Focus, Transducer 8818, 6/9 MHz).
  Biopsy cores will be numbered according to ROI number and topography. Specimens will be processed and evaluated by a genitourinary pathologist. Tumor foci will be quantified and graded according to the ISUP consensus conference on Gleason grading.

SUMMARY:
This is prospective single-arm case-control study designed to compare in parallel PSMA PET/TRUS (trans-rectal or trans-perineal) fusion biopsy ("experimental test") with mpMRI/TRUS fusion prostate biopsy ("standard test") in men with a high suspicion of PCa after at least one negative biopsy.

DETAILED DESCRIPTION:
All patients fulfilling inclusion criteria and providing informed consent to the study will undergo mpMRI and PSMA PET followed by software assisted fusion biopsy, performed in day-hospital setting.

The inclusion criteria are: blood PSA level >4.0ng/ml; free-to-total PSA ratio <20%; progressive rise of PSA levels in two consecutive blood samples despite antibiotics; serum blood tests suspicious for PCa; at least one previous negative biopsy (min 12 cores); ASAP and/or high-grade PIN; negative digital rectal examination.

The exclusion criteria are: antiandrogen therapy; prostate needle biopsy <21 days before PET and/or mpMRI; known active secondary cancer; endorectal coil/probe not applicable; active prostatitis; anaphylaxis against gadolinium-DOTA.

The total duration of the project is 36 months. We expect to enroll the first patient within 1 month after study activation, and complete recruitment within 30 months. Completion of all study analyses on biological materials and experimental imaging is expected within 32 months. The last period is planned for data analysis, biostatistics and manuscript preparation.

All patients eligible according to inclusion criteria and having signed the informed consent will undergo 68Ga-PSMA PET/CT and mpMRI scans within one month distance from each. Dedicated software for image visualization will be used to interpret and quantify 68Ga-PSMA PET/CT SUVmax and SUVratio. Images will be analyzed by an expert nuclear physician; who will proceed to the definition of the suspicious areas candidate to biopsy. mpMRI will be evaluated by an expert radiologist using the following phases: morphological, diffusion-weighted imaging (DWI) and spectroscopy. Reading criteria for mpMRI will be determined based on PI-RADS ver.2 [29]. Target delineation on PSMA PET and mpMRI will be performed as previously described [References].

Biopsy session will be completed within one month from 68Ga-PSMA PET/CT and mpMRI scans. Targeted TRUS-fusion needle biopsy will be performed for all lesions detected with PET and mpMRI. A subsequent randomized biopsy sampling consisting of 12 samples will be performed from the peripheral region of the prostate. The biopsy frustules will then be evaluated by an expert pathologist on PCa detection.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* blood PSA level >4.0ng/ml;
* free-to-total PSA ratio <20%;
* progressive rise of PSA levels in two consecutive blood samples despite antibiotics;
* serum blood tests suspicious for PCa;
* at least one previous negative biopsy (min 12 cores);
* ASAP and/or high-grade PIN;
* negative digital rectal examination.

Exclusion Criteria:

* antiandrogen therapy;
* prostate needle biopsy <21 days before PET and/or mpMRI;
* known active secondary cancer;
* endorectal coil/probe not applicable;
* active prostatitis;
* anaphylaxis against gadolinium-DOTA.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, Specificity, NPV, PPV, Accuracy | 36 months
  To evaluate the diagnostic performance of PSMA PET-TRUS fusion prostate biopsy in determining the presence of PCa in comparison to mpMRI-TRUS fusion prostate biopsy analyzed in parallel in the same subset of patients.

SECONDARY OUTCOMES:
Standardized uptake value and Gleason Score | 36 months
  To determine the correlations between the "index test" standardized uptake values (i.e. SUVmax, SUVratio; SUVmean) and the histopathological characteristics of the specimen (Gleason Score) in order to validate optimal cut-off points able to detect intraprostatic malignancy and differentiate clinically relevant PCa lesions.
Number of spared biopsies | 36 months
  To determine the clinical utility of the "index test" compared to the "standard test in terms of number of spared biopsies compared to mpMRI.
Cost-effectiveness | 36 months
  To determine the clinical utility of the "index test" compared to the "standard test in terms of cost-effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Egesta Lopci, MD, PhD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopci E, Lughezzani G, Castello A, Saita A, Colombo P, Hurle R, Peschechera R, Benetti A, Zandegiacomo S, Pasini L, Casale P, Pietro D, Bevilacqua G, Balzarini L, Buffi NM, Guazzoni G, Lazzeri M. Prospective Evaluation of 68Ga-labeled Prostate-specific Membrane Antigen Ligand Positron Emission Tomography/Computed Tomography in Primary Prostate Cancer Diagnosis. Eur Urol Focus. 2021 Jul;7(4):764-771. doi: 10.1016/j.euf.2020.03.004. Epub 2020 Apr 17. PMID 32312701
- [Background] Lopci E, Lughezzani G, Castello A, Colombo P, Casale P, Saita A, Buffi NM, Guazzoni G, Chiti A, Lazzeri M. PSMA-PET and micro-ultrasound potential in the diagnostic pathway of prostate cancer. Clin Transl Oncol. 2021 Jan;23(1):172-178. doi: 10.1007/s12094-020-02384-w. Epub 2020 May 23. PMID 32447644
- [Background] Lopci E, Saita A, Lazzeri M, Lughezzani G, Colombo P, Buffi NM, Hurle R, Marzo K, Peschechera R, Benetti A, Zandegiacomo S, Pasini L, Lista G, Cardone P, Castello A, Maffei D, Balzarini L, Chiti A, Guazzoni G, Casale P. 68Ga-PSMA Positron Emission Tomography/Computerized Tomography for Primary Diagnosis of Prostate Cancer in Men with Contraindications to or Negative Multiparametric Magnetic Resonance Imaging: A Prospective Observational Study. J Urol. 2018 Jul;200(1):95-103. doi: 10.1016/j.juro.2018.01.079. Epub 2018 Feb 1. PMID 29409824
- [Background] Lopci E, Lazzeri M. Re: Michael S. Hofman, Nathan Lawrentschuk, Roslyn J. Francis, et al. Prostate-specific Membrane Antigen PET-CT in Patients with High-risk Prostate Cancer Before Curative-intent Surgery or Radiotherapy (proPSMA): A Prospective, Randomised, Multi-centre Study. Lancet 2020;395:1208-16: PSMA Positron Emission Tomography: One Tracer Fixes Them All! Eur Urol. 2020 Sep;78(3):e131-e132. doi: 10.1016/j.eururo.2020.06.054. Epub 2020 Jul 9. No abstract available. PMID 32653324
- [Background] Lopci E, Colombo P, Lazzeri M. Mismatched Imaging Findings of Prostate Cancer Diagnosis: 68 Ga-PSMA PET/CT vs mpMRI. Nucl Med Mol Imaging. 2021 Aug;55(4):199-202. doi: 10.1007/s13139-021-00701-x. Epub 2021 Jun 2. PMID 34422131
- [Background] Lopci E, Piccardo A, Lazzeri M. Prostate cancer imaging and therapeutic alternatives with highly specific molecular 'probes'. BJU Int. 2019 Aug;124(2):188-189. doi: 10.1111/bju.14713. Epub 2019 Mar 14. No abstract available. PMID 30785658
- [Background] Lopci E, Guazzoni G, Lazzeri M. 68Ga Prostate-specific Membrane Antigen PET/CT for Primary Diagnosis of Prostate Cancer: Complementary or Alternative to Multiparametric MR Imaging. Radiology. 2018 May;287(2):725-726. doi: 10.1148/radiol.2017172607. No abstract available. PMID 29668418
- [Background] Lazzeri M, Lopci E, Lughezzani G, Colombo P, Casale P, Hurle R, Saita A, Leonardi L, Lista G, Peschechera R, Pasini L, Rodari M, Zandegiacomo S, Benetti A, Cardone P, Mrakic F, Balzarini L, Chiti A, Guazzoni G, Buffi NM. Targeted 11C-choline PET-CT/TRUS software fusion-guided prostate biopsy in men with persistently elevated PSA and negative mpMRI after previous negative biopsy. Eur J Hybrid Imaging. 2017;1(1):9. doi: 10.1186/s41824-017-0011-1. Epub 2017 Nov 1. PMID 29782590
- [Background] Evangelista L, Lopci E. Re: Hendrik Van Poppel, Renee Hogenhout, Peter Albers, et al. Early Detection of Prostate Cancer in 2020 and Beyond: Facts and Recommendations for the European Union and the European Commission. Eur Urol 2021;79:327-9: Early Detection of Prostate Cancer in High-risk Patients with Negative Fusion Biopsy. Eur Urol. 2021 Jul;80(1):e24-e27. doi: 10.1016/j.eururo.2021.04.026. Epub 2021 May 2. No abstract available. PMID 33947593